CLINICAL TRIAL: NCT07209202
Title: Fructose Metabolism Effects on the Liver: Unraveling the Role of Defective Intestinal GNG in Individuals With Obesity
Brief Title: Fructose Intestinal Gluconeogenesis
Acronym: FIG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Touro University, California (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jean-marc Schwarz, Professor, Touro University, California
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: M-2624; R01DK140477 (NIH)
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants; Obese But Otherwise Healthy Participants
Keywords: Fructose; Sugar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High fructose meals, oral 13C fructose (Experimental): Liquid meals will be fed, containing 55% total carbohydrate (16% fructose), 30% fat, 15% protein, and a tracer amount of 13C fructose.
  Interventions: Other: High fructose meal; Other: 13C labeled fructose, oral
- High Fructose Meals, IV 13C Fructose (Experimental): Liquid meals will be fed, containing 55% total carbohydrate (16% fructose), 30% fat, 15% protein. A tracer amount of 13C fructose will be administered intravenously.
  Interventions: Other: High fructose meal; Other: 13C labeled fructose, intravenous
- Low fructose meals, oral fructose tracer (Experimental): Liquid meals will be fed, containing 55% total carbohydrate (6% fructose), 30% fat, 15% protein, and a tracer amount of 13C fructose.
  Interventions: Other: Low fructose meal; Other: 13C labeled fructose, oral
- Low fructose meals, IV 13C fructose tracer (Experimental): Liquid meals will be fed, containing 55% total carbohydrate (6% fructose), 30% fat, 15% protein. A tracer amount of 13C fructose will be administered intravenously.
  Interventions: Other: Low fructose meal; Other: 13C labeled fructose, intravenous

INTERVENTIONS:
Other: High fructose meal — Liquid meals containing 55% total carbohydrate (16% fructose), 30% fat, 15% protein.
  Arms: High Fructose Meals, IV 13C Fructose; High fructose meals, oral 13C fructose
Other: Low fructose meal — 55% total carbohydrate (6% fructose), 30% fat, 15% protein.
  Arms: Low fructose meals, IV 13C fructose tracer; Low fructose meals, oral fructose tracer
Other: 13C labeled fructose, oral — Tracer amount of 13C labeled fructose administered orally in the meals.
  Arms: High fructose meals, oral 13C fructose; Low fructose meals, oral fructose tracer
Other: 13C labeled fructose, intravenous — Tracer amount of 13C fructose administered intravenously
  Arms: High Fructose Meals, IV 13C Fructose; Low fructose meals, IV 13C fructose tracer

SUMMARY:
This study will test the hypothesis that within a defined range of fructose intake, the ability to convert fructose to glucose (via gluconeogenesis) in the small intestine plays a protective role for the liver, shielding it from the deleterious effects of fructose. We will investigate whether this protective effect of the intestine is impaired in individuals with obesity.

DETAILED DESCRIPTION:
Qualified participants will undergo a sugar tolerance test at baseline and then randomized to undergo four separate outpatient tracer/feeding studies in a crossover fashion. After an overnight fast, a six-hour fed tracer study will be initiated, during which participants will consume liquid meals containing stable isotopes at regular intervals and receive other isotopes intravenously. Meal composition will differ only by fructose content (High vs. Low) and tracer (oral vs. intravenous 13C-labeled fructose). Blood and urine samples will be collected frequently throughout the study. Each visit will be performed approximately three weeks apart. Vital signs and anthropometrics will be measured at each clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30 to 38 kg/m2 (obese group) or BMI 19 to 25 kg/m2 (lean group)

Exclusion Criteria:

* Pregnancy or lactation within the past six months;
* Type 1 or 2 diabetes mellitus (including fasting glucose ≥126 mg/dL, HgbA1c ≥6.5%);
* History of liver disease or AST and ALT 2x above the upper limit of normal;
* Fasting triglyceride > 300 mg/dl; total cholesterol levels above the 95th percentile for age and sex;
* Hemoglobin (Hgb) <12.5g/d or hematocrit<3x Hgb value;
* Report of HIV or hepatitis B or C infection;
* History of cancer, other than basal cell or squamous cell carcinoma or kidney disease stage 3 or higher or patients currently on dialysis;
* Use of any anti-diabetic medications or hypolipidemic agents in the past six months;
* History of surgical procedure for obesity;
* Change in body weight >5% in the past six months (by self-report);
* History of other conditions known to affect insulin sensitivity and lipid metabolism (e.g., polycystic ovary syndrome), history of galactosemia, hereditary fructose intolerance, or who test positive for fructose malabsorption at screening;
* Known intolerance to acetaminophen.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Fru-GNG | 6 hours
  Total amount of fructose converted to glucose
Fru-hGNG | 6 hours
  Amount of fructose converted to glucose in the liver
Fru-iGNG | 6 hours
  Amount of fructose converted to glucose in the intestine
De novo lipogenesis (DNL) | 6 hours
  Percent of newly synthesized palmitate

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Schwarz, PhD, Principal Investigator — Touro University, California; Grace M Jones, PhD, Principal Investigator — Touro University, California

IPD SHARING:
Plan to Share IPD: Yes
The de-identified clinical and laboratory data set will be made available upon request to academic investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data will be made available for at least 5 years from publication of the primary manuscript.
Access Criteria: Academic investigators may request data and supporting information upon request to the PI.